CLINICAL TRIAL: NCT04156607
Title: The Effects of Kinesiotaping on Balance in Children With Down Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, pelin atalan, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/05-23
Record Dates: First submitted 2019-10-29; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Down Syndrome; Balance
Keywords: Down Syndrome; Postural Balance; Kinesio Taping
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: The study was carried out with the participation of 3 groups as kinesio taping application group with Down Sydnrome children (KT) (n=12, DS), sham taping application group with Down Syndrome children (ST) (n=12, DS) and healthy control with healty children (HC) (n=12). Healty children took no taping applications. KT group took Kinesio tape, ST group took sham taping evaluated 2 times after the tapings (immediately and 45 minutes later).
Who Masked: Participant
Masking Description: Half of the children with DS (Sham taping group) took sham taping application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio taping group (KT) (Experimental): Kinesio taping applied to plantar soles of these children with Down Syndrome. Epidermis-Dermis-Fascia technique was used for providing sensory input from soles.
  The application was performed on both feet.
  Interventions: Other: Kinesio taping
- Sham taping group (ST) (Sham Comparator): A random taping was performed using Kinesio tape but without using Kinesiotaping techniques for sham taping. The application was performed on both feet
  Interventions: Other: Sham taping
- Healty control group (No Intervention): This group took no intervention but all balance assessments once.

INTERVENTIONS:
Other: Kinesio taping — For the fascia technique, one part of the band which were divided by 4 fans is adhered on Achilles tendon to the heel with a 0% stretch. Then the plantar fascia was stretched by the examiner and the toes were extended (ankle dorsiflexion, toe extension) and the divided part of the band was applied toward the metatarsal heads with paper-off technique (5-15%).
  Arms: Kinesio taping group (KT)
Other: Sham taping — ''I'' bant were cut from the middle point of the Achilles tendon to the metatarsal heads. The band was applied from the Achilles tendon to the metatarsal heads without any stretching of plantar fascia and band.
  Arms: Sham taping group (ST)

SUMMARY:
This study aimed to explore the effects of Kinesio tape applied to plantar soles on balance in children with Down Syndrome (DS). Two groups including children with DS and a group with their typically developing peers evaluated. Half of the children with DS took Kinesio tape application to the plantar soles and the other half took sham taping application. All children evaluated with dynamic and static balance measurements and DS children evaluated immediately after taping and 45 minutes after taping again with the same measurements.

DETAILED DESCRIPTION:
Balance is one of the most problematic issues in children with DS. Mechanoreceptors of plantar region of the foot helps to regulate human erect posture and balance. Studies shows that inputs from foot sole give a positive effect in improving balance both in healthy and neurologically demaged subjects. Kinesio tape is a supportive method in physiotherapy with it's proprioceptive input giving effects. It is aimed to show the acute effects of Kinesio tape on balance parameters in children with DS.

ELIGIBILITY:
The inclusion criteria for healthy children:

* Not having any orthopedic or neurological disorder
* To understand and do the commands given
* Being willing to participate in the study

The inclusion criteria for children with DS:

* To have diagnosis of DS
* Not having any orthopedic or neurological disorder in addition the DS
* To understand and do the commands given
* Being willing to participate in the study.

Exclusion criteria for all children:

* Auditory and visual problems (not using glasses)
* Operated in last 6 months prior to he study

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Static balance | Static balance evaluated with Modified Clinical test of Sensory Interaction on Balance (MCTSIB) for Down syndrome children before the randomization and taping application. The healthy control group took this test once. This test takes 1-2 minutes.
  Static balance is the ability to keep the body upward without falling when the person is not moving.
Functional (dynamic) balance | Dynamic balance evaluated with Timed Up and Go for Down syndrome children before the randomization and taping application. The healthy control group took this test once. This test takes 1-2 minutes.
  Dynamic balance is the ability to keep the body upward without falling when the person is moving and in challenging conditions like walking, running, jumping, reaching etc.
Static balance | Static balance evaluated with Modified Clinical test of Sensory Interaction on Balance (MCTSIB) for Down syndrome children immediately after the taping application. This test takes 1-2 minutes.
  Static balance is the ability to keep the body upward without falling when the person is not moving.
Functional (dynamic) balance | Dynamic balance evaluated with Timed Up and Go test for Down syndrome children immediately after the taping application. This test takes 1-2 minutes.
  Dynamic balance is the ability to keep the body upward without falling when the person is moving and in challenging conditions like walking, running, jumping, reaching etc.
Static balance | Static balance evaluated with Modified Clinical test of Sensory Interaction on Balance (MCTSIB) for Down syndrome children 45 minutes after the taping application. This test takes 1-2 minutes.
  Static balance is the ability to keep the body upward without falling when the person is not moving.
Functional (dynamic) balance | Dynamic balance evaluated with Timed Up and Go test for Down syndrome children 45 minutes after the taping application. This test takes 1-2 minutes.
  Dynamic balance is the ability to keep the body upward without falling when the person is moving and in challenging conditions like walking, running, jumping, reaching etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylül University, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alsakhawi RS, Elshafey MA. Effect of Core Stability Exercises and Treadmill Training on Balance in Children with Down Syndrome: Randomized Controlled Trial. Adv Ther. 2019 Sep;36(9):2364-2373. doi: 10.1007/s12325-019-01024-2. Epub 2019 Jul 12. PMID 31301057
- [Background] Kavounoudias A, Roll R, Roll JP. Foot sole and ankle muscle inputs contribute jointly to human erect posture regulation. J Physiol. 2001 May 1;532(Pt 3):869-78. doi: 10.1111/j.1469-7793.2001.0869e.x. PMID 11313452
- [Background] Tutun Yumin E, Simsek TT, Sertel M, Ankarali H, Yumin M. The effect of foot plantar massage on balance and functional reach in patients with type II diabetes. Physiother Theory Pract. 2017 Feb;33(2):115-123. doi: 10.1080/09593985.2016.1271849. Epub 2017 Jan 17. PMID 28095093
- [Background] Hu Y, Zhong D, Xiao Q, Chen Q, Li J, Jin R. Kinesio Taping for Balance Function after Stroke: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2019 Jul 16;2019:8470235. doi: 10.1155/2019/8470235. eCollection 2019. PMID 31379969